CLINICAL TRIAL: NCT00608894
Title: A Phase II, Open-Label, Multi-Center, Prospective, Randomized Study of LCP-Tacro Tablets vs. Azathioprine, in Combination With Corticosteroids, for the Treatment of Autoimmune Hepatitis
Brief Title: LCP-Tacro vs. Azathioprine for the Treatment of Autoimmune Hepatitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was discontinued due to slow enrollment
Sponsor: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCP-Tacro Study 2016
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune hepatitis; Chronic active hepatitis
MeSH Terms: conditions — Hepatitis, Autoimmune; Hepatitis, Chronic | interventions — Tacrolimus; Azathioprine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LCP-Tacro (Experimental): LCP-Tacro tablets(1,2,and 5mg tacrolimus)+ prednisone tablets(5mg)
  Interventions: Drug: LCP-Tacro (tacrolimus)
- Azathioprine (Active Comparator): Azathioprine tablets(50mg)+ prednisone tablets(5mg)
  Interventions: Drug: Azathioprine

INTERVENTIONS:
Drug: LCP-Tacro (tacrolimus) — LCP-Tacro(tacrolimus)tablets starting at 2 mg once daily, then adjusted to achieve and maintain target whole blood tacrolimus levels of 3 - 6 ng/mL, plus prednisone 30 mg/day for one week, then 20 mg/day for one week, then 15 mg/day for two weeks, then 10 mg/day through Month 6.
  Other Names: 1,2,and 5mg tacrolimus tablets
  Arms: LCP-Tacro
Drug: Azathioprine — Azathioprine tablets 50 - 100 mg (approximately 1 mg/kg) once daily, plus prednisone 30 mg/day for one week, then 20 mg/day for one week, then 15 mg/day for two weeks, then 10 mg/day through Month 6.
  Other Names: 50mg azathioprine tablets + 5mg prednisone tablets
  Arms: Azathioprine

SUMMARY:
An open-label, multi-center, prospective, randomized study to evaluate the efficacy, safety and tolerability of LCP-Tacro tablets given once daily vs. azathioprine, each in combination with prednisone, for the treatment of autoimmune hepatitis (AIH).

DETAILED DESCRIPTION:
An open-label, multi-center, prospective, randomized study to evaluate the efficacy, safety and tolerability of LCP-Tacro tablets given once daily vs. azathioprine for the treatment of autoimmune hepatitis (AIH).

Patients with histologically confirmed chronic hepatitis who fulfill criteria established by the International Autoimmune Hepatitis Group (IAIHG) and Inclusion and Exclusion criteria will be enrolled after having signed an informed consent document.

Up to 60 patients will be randomized (1:1) to receive treatment with LCP-Tacro + prednisone vs. azathioprine (AZA) + prednisone.

* LCP-Tacro will be started at 2 mg once daily (q.d.) with weekly measurement of tacrolimus whole blood trough levels and adjustment of the daily dose of LCP-Tacro to achieve target tacrolimus levels of 3 - 6 ng/mL. Patients with histological evidence of cirrhosis and a Model for End-Stage Liver Disease (MELD) score ≤ 8 will commence LCP-Tacro at a fixed dose of 1 mg once daily, with subsequent dosage adjustments to maintain tacrolimus trough levels at 3 - 6 ng/mL.
* AZA will be started at 50 - 100 mg (approximately 1 mg/kg) once daily (q.d.).

Patients will also commence treatment with prednisone 30 mg/day for one week, then 20 mg/day for one week, then 15 mg/day for two weeks, then 10 mg/day through Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Men and women at least 18 years of age with a diagnosis of definite or probable AIH defined by the revised International Autoimmune Hepatitis Group (IAIHG) criteria
* Elevation of serum ALT ≥ 1.5 times the upper limit of normal
* Liver biopsy showing chronic hepatitis consistent with AIH
* Patients able to swallow the study medication
* Patients capable of understanding the purposes and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study
* Women of childbearing potential must have a negative serum pregnancy test within seven days prior to receiving study medication and agree to use contraceptive measures to avoid pregnancy during participation in the trial.

Exclusion Criteria:

* Patients with other concurrent liver disease
* Patients with cirrhosis on liver biopsy with a MELD score > 15
* Patients with a history or presence of decompensated liver disease
* Patients with serum creatinine ≥ 1.5 mg/dL prior to enrollment
* Patients positive for HCV RNA or Hepatitis B surface antigen (HBsAg)
* Patients with a history of alcohol intake > 25 g/day within the past six months
* Patients with TSH outside normal range accompanied by an abnormal T4
* Patients with alpha-fetoprotein ≥ 20 ng/mL
* Patients with severe anemia (hemoglobin < 8 g/dL), leukopenia (WBC < 4000/mm3), or thrombocytopenia (platelet count < 100,000/mm3)
* Patients with a history of recent exposure to hepatotoxic drugs
* Patients who require therapy with any immunosuppressive agent other than those prescribed in the study
* Patients unable or unwilling to provide informed consent
* Pregnant or nursing women
* Patients with reproductive potential who are unwilling/unable to use a double barrier method of contraception
* Patients who have been treated with another investigational agent in the three months prior to enrollment
* Patients receiving any drug interfering with tacrolimus metabolism
* Patients with current malignancy or a history of malignancy (within the past 5 years), except basal or non-metastatic squamous cell carcinoma of the skin that has been treated successfully
* Patients with uncontrolled concomitant infection, a systemic infection requiring treatment, or any other unstable medical condition that could interfere with the study objectives
* Patients with severe diarrhea, vomiting, active peptic ulcer or gastrointestinal disorder that may affect the absorption of tacrolimus
* Patients with a known hypersensitivity to azathioprine, corticosteroids or tacrolimus
* Patients with any form of current substance abuse, psychiatric disorder or a condition that, in the opinion of the Investigator, may invalidate communication with the Investigator
* Patients who are recipients of an organ transplant or who require treatment with immunosuppressives or corticosteroids for any disease other than AIH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Y Minuk, M.D., Principal Investigator — University of Manitoba Health Sciences Centre, Winnipeg; Andrew Mason, MD, Principal Investigator — University of Alberta, Edmonton; Russell H Wiesner, MD, Principal Investigator — Mayo Clinic, Rochester, MN; John M Vierling, MD, Principal Investigator — Baylor College of Medicine; Velimir A Luketic, MD, Principal Investigator — Virginia Commonwealth University, Richmond, VA; Joseph A Odin, MD, PhD, Principal Investigator — Mount Sinai Medical Center, New York, NY; Elizabeth Carey, MD, Principal Investigator — Mayo Clinic; John R Lake, MD, Principal Investigator — University of Minnesota; Barry G Rosser, MD, Principal Investigator — Mayo Clinic; Steven L Flamm, MD, Principal Investigator — Northwestern University; Kevork M Peltekian, MD, Principal Investigator — Queen Elizabeth II Health Sciences Centre; Mark G Swain, MD, Principal Investigator — University of Calgary
Locations (12):
- United States (8):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - St. Luke's Advanced Liver Therapies, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Canada (4):
  - Heritage Medical Research Clinic, Calgary, Alberta
  - Zeildler Ledcor Centre, Edmonton, Alberta
  - John Buhler Research Centre, University of Manitoba Health Sciences Centre, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCP-Tacro | Azathioprine
Started | 7 | 6
Completed | 7 | 4 (One patient was granted permission to crossover to LCP-Tacro due to treatment intolerance)
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCP-Tacro | Azathioprine | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Median (Full Range); unit: years] | 50 [19 to 70] | 56 [47 to 65] | 53 [19 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 6 | 6 | 12
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Remission of (AIH) at Month 6.
Description: Percent of patients that achieve biochemical remission of (AIH) at Month 6 during treatment with LCP-Tacro + prednisone or azathioprine + prednisone. Biochemical remission is defined as ALT, total bilirubin and gamma globulin within normal limits.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | LCP-Tacro | Azathioprine
Number analyzed (Participants) | 7 | 6
Participants | 3 | 4

2. Secondary Outcome: Biochemical Remission by Month 3.
Description: Percent of patients who achieve biochemical remission by Month 3 during treatment with LCP-Tacro + prednisone or azathioprine + prednisone. Biochemical remission is defined as ALT, total bilirubin and gamma globulin within normal limits.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | LCP-Tacro | Azathioprine
Number analyzed (Participants) | 7 | 4
Participants | 2 | 4

3. Secondary Outcome: Incomplete Response, Treatment Failure, or a Case of Relapse at 6 Months
Description: Percents of patients in each treatment group classified as having an incomplete response (defined as some or no improvement during therapy), a treatment failure (defined as permanent discontinuation of the regimen originally randomized to), or a case of relapse (recurrence following achievement of remission)
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- LCP-Tacro: LCP-Tacro tablets(1,2,and 5mg tacrolimus)+ prednisone tablets(5mg)
  LCP-Tacro (tacrolimus): LCP-Tacro(tacrolimus)tablets starting at 2 mg once daily, then adjusted to achieve and maintain target whole blood tacrolimus levels of 3 - 6 ng/mL, plus prednisone 30 mg/day for one week, then 20 mg/day for one week, then 15 mg/day for two weeks, then 10 mg/day through Month 6.
  Seven patients were randomized to LCP-Tacro. All 7 (100%) completed the study and no crossovers or early withdrawals occurred.
- Azathioprine: Azathioprine tablets(50mg)+ prednisone tablets(5mg)
  Azathioprine: Azathioprine tablets 50 - 100 mg (approximately 1 mg/kg) once daily, plus prednisone 30 mg/day for one week, then 20 mg/day for one week, then 15 mg/day for two weeks, then 10 mg/day through Month 6.
  Six patients were randomized to Azathioprine. One patient (16.7%) was granted permission to crossover to LCP-Tacro due to treatment intolerance. Two patients (33.3%) withdrew early, and 4 patients (66.7%) completed the study.
Arm/Group | LCP-Tacro | Azathioprine
Number analyzed (Participants) | 7 | 6
Participants
  Incomplete response | 4 | 1
  Treatment failure | 0 | 1
  Relapse | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: One patient (AZA) crossed over to treatment with LCP - Tacro after 8 weeks of treatment and is included in the original treatment group to which he was randomized (AZA)
Arm/Group | LCP-Tacro | Azathioprine
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 6/7 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCP-Tacro (N=7) | Azathioprine (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 2
Headache (Nervous system disorders) | 2 | 0
Tremor (Nervous system disorders) | 2 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
The study was discontinued due to slow enrollment. Consequently, the number of patients enrolled in the study was too small to permit meaningful statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study is a multicenter collaborative investigation and the clinical trial results are to be published as a collaborative manuscript. Authorship will reflect varying levels of individual contribution to the study by the individual PI's.